CLINICAL TRIAL: NCT06808230
Title: Cocoa Flavanols for Migraine: A Pilot Study
Brief Title: Cocoa Extract for Migraine Trial
Acronym: CORAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Pamela M. Rist, ScD, Associate Epidemiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2024P003655; U01AT012611 (NIH)
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Migraine
Keywords: migraine; cocoa extract; cocoa flavanol
MeSH Terms: conditions — Migraine Disorders | interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants assigned to this arm will take four placebo pills per day.
  Interventions: Dietary Supplement: Cocoa extract placebo
- 500 mg cocoa extract (Experimental): Participants assigned to this arm will take two 250 mg cocoa extract pills per day and two placebo pills per day
  Interventions: Dietary Supplement: Cocoa extract
- 1000 mg cocoa extract (Experimental): Participants assigned to this arm will take four 250 mg cocoa extract pills per day
  Interventions: Dietary Supplement: Cocoa extract

INTERVENTIONS:
Dietary Supplement: Cocoa extract — Cocoa extract manufactured as 250 mg capsules
  Arms: 1000 mg cocoa extract; 500 mg cocoa extract
Dietary Supplement: Cocoa extract placebo — Cocoa extract placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the feasibility of recruitment and adherence to a high-dose cocoa extract supplement in individuals diagnosed with episodic migraine. The main questions it aims to answer are:

* Will we be able to enroll 114 participants during the recruitment period?
* Will participants take study pills daily during the pill-taking period?

Researchers will compare two doses of cocoa extract to placebo to determine the acceptability of higher doses of cocoa extract supplementation in this patient population.

Participants will be asked to:

* Provide two urine samples
* Complete daily questionnaires
* Take four study pills a day for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged ≥18 years
* Self-reported clinician diagnosis of migraine with or without aura which does not meet criteria for chronic migraine (according to the International Classification of Headache Disorders 3rd edition)

  * Individuals with self-reported migraine will need to report a clinician diagnosis of migraine and be classified as having migraine or probable migraine by the American Migraine Study (AMS) migraine screener. The AMS migraine screener, which has a sensitivity of 100% and a specificity of 82% for the diagnosis of migraine will be used to confirm self-reported migraine status.
  * History of migraine dating for at least one year
* Self-report of 4 to 14 migraine attacks during the 30 days prior to enrollment in the study
* Completion of at least 22 headache diary days during the 28 day run-in period

  o Report migraine frequency between 4 to 14 days during the 28 day run-in period
* If currently using medications to prevent or treat migraine, no new medication use within the past 3 months
* No new use of behavioral interventions within the past 3 months and/or agree to not begin new behavioral interventions during this trial
* Be willing to complete all study procedures and be randomized to all interventional groups
* Be fluent in English
* Own an iPhone or Android device and be willing to download MyCap to the device

Exclusion Criteria:

* Self-reported history of stroke or transient ischemic attack; history of brain surgery or spine surgery; currently receiving treatment for a concussion; and self-reported diagnosis of cluster headache, brain tumor, brain aneurysm, traumatic brain injury, multiple sclerosis, epilepsy, schizophrenia, or bipolar disorder
* Kidney failure or current dialysis treatment or any medical condition which the participant believes could lead to difficulty complying with the protocol
* Current alcohol or substance abuse (self-reported)
* Self-reported clinician diagnosis of medication overuse headache
* Currently or recently (past 6 months) received Botox treatment for migraine
* Failure to return the baseline urine sample
* Currently pregnant, nursing, or intending to become pregnant during the study period.
* Unwilling to forgo use of out-of-study supplements of cocoa extract during the trial
* Extreme sensitivity to caffeine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 15 months
  We will be able to recruit and randomize 114 eligible individuals
Retention | From run-in to end of treatment at 12 weeks
  Retention will be quantified by the proportion of subjects who record their migraines for at least 22 out of 28 days during run-in and the last four weeks of the intervention and complete all questionnaires at baseline and follow-up
Adherence | 12 week intervention period
  Adherence will be calculated as the proportion of participants who miss no more than 12 days of study pills (i.e. participants will consume study pills on 85% of the intervention days)

SECONDARY OUTCOMES:
Migraine days | Four week run-in period and final four weeks of the 12 week intervention period
  Number of migraine attacks as recorded in migraine diaries
Responder rate | Four week run-in period and final four weeks of the 12 week intervention period
  Proportion of individuals who experience a ≥50% reduction in migraine days
Migraine severity | Four week run-in period and final four weeks of the 12 week intervention period
  Four-point scale with categories of "absent, mild, moderate, or severe".
Adverse events | 12 week intervention period
  Potential side effects and adverse events
Reports of worsening of migraine symptoms | 12 week intervention period
  Worsening of photophobia, phonophobia, or osmophobia, and worsening of aura symptoms in the past week compared to the week prior
Allodynia Symptom Checklist | Baseline and end of the 12 week intervention period
  Survey assessing how often individuals with migraine experience allodynia
Headache Related Disability (HIT-6) | Baseline and end of the 12 week intervention period
  Evaluates the impact headaches have on a patient's life and
PROMIS-29 | Baseline and end of the 12 week intervention period
  Measures of patient-reported health status for physical, mental, and social well-being
Urine levels of gamma-valerolactone metabolites (gVLM) | Four week run-in period and final four weeks of the 12 week intervention period
  Biomarker of dietary flavanol intake

CONTACTS AND LOCATIONS:
Overall Officials: Pamela M Rist, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Cleaned, item-level spreadsheet data for all variables will be shared openly, along with example quantifications and transformations from initial raw data
Supporting Information: Analytic Code
Time Frame: Data will be shared no later than time of the final publication of study results or the end of the performance period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 10 years after the end of the funding period.
Access Criteria: Data and supporting materials will be shared on the Harvard Dataverse. The data that is shared will be shared by unrestricted download.